CLINICAL TRIAL: NCT01432301
Title: An Open-Label Protocol for the Use of Uridine Triacetate as an Antidote to Treat Patients at Excess Risk of 5-Fluorouracil Toxicity Due to Overdosage or Impaired Elimination
Brief Title: Uridine Triacetate as Antidote for Patients at Excess Risk of 5-FU Toxicity Due to Overdosage or Impaired Elimination
Status: Approved for marketing | Type: Expanded Access
Sponsor: Wellstat Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 401.10.001
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Toxicity Due to Chemotherapy
Keywords: fluorouracil overdose; fluorouracil toxicity; capecitabine overdose; capecitabine toxicity
MeSH Terms: interventions — uridine triacetate

INTERVENTIONS:
Drug: uridine triacetate — uridine triacetate granules, 10gms, q6H x 20 doses
  Other Names: PN401; Vistogard

SUMMARY:
The purpose of this study is to provide emergency treatment of adult and pediatric patients:

* Following a fluorouracil or capecitabine overdose regardless of the presence of symptoms or
* Who exhibit early-onset, severe or life-threatening toxicity affecting the cardiac or central nervous systems, and/or early-onset, unusually severe adverse reactions (e.g., gastrointestinal toxicity and/or neutropenia) within 96 hours following the end of fluorouracil or capecitabine administration.

DETAILED DESCRIPTION:
Demographics, baseline disease information, prior disease-directed therapy including fluorouracil or capecitabine, and details of the fluorouracil or capecitabine overexposure (dose, cause, and timing) will be collected. Adverse events information will be collected and recorded. Patients will be followed for 30 days unless the patient expires or resumes chemotherapy within the 30 day period.

ELIGIBILITY:
Inclusion Criteria:

* The patient received a fluorouracil or capecitabine overdose (regardless of the presence of symptoms) or
* The patient is exhibiting early-onset, severe or life-threatening toxicity affecting the cardiac or central nervous system, and/or early-onset, unusually severe adverse reactions (e.g., gastrointestinal toxicity and/or neutropenia) within 96 hours following the end of fluorouracil or capecitabine administration
* Judged by the Investigator to have the initiative and means to be compliant with the protocol
* Able to take oral medications
* Able to start treatment with uridine triacetate within 96 hours after the end of fluorouracil or capecitabine administration
* Provides written informed consent (patient or legally authorized representative)

Exclusion Criteria:

* Has a known allergy to uridine triacetate or any of its excipients
* Unable to have the initiative and means to be compliant with the protocol
* Unable to be compliant with taking oral medications
* More than 96 hours have elapsed since the completion of 5-FU dosing
* Unable to provide written informed consent (patient or legally authorized representative)

Sex: All
Age Groups: Child, Adult, Older Adult